CLINICAL TRIAL: NCT03487328
Title: A New Technique for Sacrospinous-Sacrotuberous Fixation for the Treatment of Uterovaginal and Vaginal Vault Prolapse: A Randomized Controlled Trial
Brief Title: A New Technique for Sacrospinous-Sacrotuberous Fixation for the Treatment of Uterovaginal and Vaginal Vault Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1729
Record Dates: First submitted 2018-03-21; First posted 2018-04-04 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Uterovaginal and Vaginal Vault Prolapse
Keywords: treatment
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified technique for Sacrospinous-Sacrotuberous Fixation (Active Comparator): Modified technique for Sacrospinous-Sacrotuberous Fixation
  Interventions: Procedure: Sacrospinous-Sacrotuberous fixation
- Conventional technique for Sacrospinous-Sacrotuberous Fixation (Active Comparator): Modified technique for Sacrospinous-Sacrotuberous Fixation
  Interventions: Procedure: Sacrospinous-Sacrotuberous fixation

INTERVENTIONS:
Procedure: Sacrospinous-Sacrotuberous fixation — Sacrospinous-Sacrotuberous fixation

SUMMARY:
This prospective interventional randomized controlled trial is conducted to compare a new technique for Sacrospinous-Sacrotuberous fixation with the traditional sacrospinous ligament fixation technique for treatment of uterovaginal and vaginal vault prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 40 to 60 years.
2. POP Q stage III & IV
3. Uterovaginal prolapse.
4. Vaginal vault prolapse.
5. BMI >35.

Exclusion Criteria:

1. Age > 40 years or < 60 years.
2. POP Q stage I or II.
3. BMI < 35.
4. Previous repair of uterovaginal or vaginal vault prolapse.
5. Comorbidity with Stress Urinary Incontinence.
6. Presence of persistent risk factor increasing intra-abdominal pressure e.g. chronic chest conditions.
7. Any significant comorbidity or psychiatric disorder that would compromise patient's consent.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with recurrence of uterovaginal and vaginal vault prolapse | 1 year

SECONDARY OUTCOMES:
blood loss | intraoperative
Injury to surrounding structures | intraoperative
  Number of participants that experience injury of important surrounding structure intraoperative
operative time | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt